CLINICAL TRIAL: NCT01879150
Title: Single Center, Open-label, Single Arm, Study Designed to Evaluate Safety, Tolerability and Efficacy of CyclaPlex Implant and Tools for Correction of First Inter-metatarsal Angle in Subjects Suffering From Hallux Valgus Deformity
Brief Title: Pilot Study of CyclaPlex Implant, an Enhanced Suture and Button Implant Device in Hallux Valgus Deformity
Acronym: CO001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mmc-cyclaplex001-il
Record Dates: First submitted 2012-09-02; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CYCLAPLEX bone anchors (Experimental): Following a 28-day screening period, eligible subjects requiring surgical correction for HV deformity (1st IMA >12degree, =<20 degree) will be enrolled to undergo HV deformity correction procedure with CYCLAPLEX under local or spinal anesthesia.
  The device is implanted via small holes drilled in 1st and 2nd metatarsals. Complementary normal medical procedures such as bunionectomy, soft tissue release and HV angle correction will be performed as required.
  Subjects will be followed-up for 50 weeks post-procedure.
  Interventions: Device: Cyclaplex bone anchor

INTERVENTIONS:
Device: Cyclaplex bone anchor — Device implantation

SUMMARY:
Single center, open-label, single arm, pilot study designed to evaluate safety, tolerability and efficacy of CYCLAPLEX device, a minimal invasive enhanced suture and button implant and surgery tools for correction of inter-metatarsal angle in subjects suffering from mild to moderate Hallux Valgus deformity

DETAILED DESCRIPTION:
INVESTIGATIONAL THERAPY Cycla Orthopedics Ltd has developed the CYCLAPLEX , a minimally invasive enhanced type of Suture and Button implant. It is intended to: (a) reduce the intermetatarsal angle (IMA) between 1MT and 2MT without osteotomy osteotomy b) reduce the risk of 2MT fractures (d) perform the implantation procedure in an easy and safe way.

The CYCLAPLEX predicated device is the "Suture and Button" type MiniTightrope. It is based on Mini Tightrope clinical experience, however with additional features to increase safety and functionality.

The CyclaPlex device comprise of two bone holders ('Anchors ') connected by a metal cord. The cord is connected to the buttons by crimp method as part of the surgery procedures The bone holders are T shape screws that are screwed into the bones after drilling holes across the 2 metatarsals. The gap in the bone as a result of the drilling is filled by the enhanced T shape buttons (screws). A nut is residing internally as part of the 1st met anchor structure. The IMA is reduced using specially designed tensioning tool CyclaPlex device is indicated for reducing intermetatarsal angles in cases where IMA is less than 200 eliminating the need for the traditional 1st metatarsal osteotomy. It used in conjunction with traditional release of the lateral MTP joint capsular structures and removal of the medial eminence as well as regular HVA reduction procedures such as AKIN.

The 2nd Metatarsal fracture risk is reduced due multiple/ accumulated factors:

(i) The hole drilled at 2nd metatarsal had been reduced significantly (ii) The hole is filled by conical screw and head. This firm anchoring method enable to distribute the horizontal forces applied during gate.

(iii) The metal screw type device enables bone growth over it and strengthen the bone at that area.

(iv) The connecting cord is housed inside the screw and has no direct touch with the bone, in both, 2nd and 1st metatarsals.

The device is delivered sterilized ( steam sterilization) double bag residing in cardboard box.

Dedicated assistive tools for multiple use are provided as well housed in a special tray intended for surgery room steam sterilization. The tools comprise of Aiming Drilling Guide,, screw driver for anchors insertion, Tensioning tool for reduction of the IMA, Crimping tool, cutter, single use drill bits

ELIGIBILITY:
Inclusion Criteria

* Adult males and female subjects, aged 20 to 75 years old, inclusive, at screening visit
* Subject weighing <100 kg and body mass index (BMI) <32 kg/m2
* Subjects with confirm diagnosis of HV deformity based on radiography assessment of IMA > 12 º and less or equal to 20degree.
* Subjects who would need osteotomy of the 1st MT as part of their surgery.
* Able and willing to comply with the requirements of the protocol.
* Able to understand and sign written informed consent to participate in the study

Exclusion criteria

* Contraindication to implantation procedure
* History of: Diabetes mellitus,Claudication vascular disease or known Peripheral Vascular Disease,Rheumatoid disease no palpable pulse (DP or PT),- Gout or any systemic inflammatory arthropathy,Osteoarthritis of first metatarsal,Neurological conditions associated with spasticity,No prior operation at 1st and 2nd Metatarsals
* Osteoporosis
* Secondary metatarsal complications including:Fracture (past or present), Aseptic necrosis or any deformity of 2nd MTH,Subject currently enrolled in or has not yet completed at least 30 days since ending
* Any condition that may jeopardize study participation (e.g. abnormal clinical or laboratory finding), the interpretation of study results or may impede the ability to obtain informed consent (e.g., mental condition)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-02 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects with 1st IMA ≤9º or reduction of more than 7º in the 1st IMA compared to Base line at last observed value (LOV). | 6 months follow up and 12 months follow up

SECONDARY OUTCOMES:
General Improvement as assessed by American Orthopaedic Foot and Ankle Society Hallux Metatarsophalangeal-lnterphalangeal Scale (AOFAS HMIS) score | 6 months, 12 months
  The AOFAS score results at each visit will be evaluated and compared to other known studies published
Pain and Functional assessment [Foot Function Index (FFI)] | 6 months 12 months
  Pain and functional index will be assesed for complete results and separately for pain and functionality
Time to full weight bear, to use of regular shoes and fashion shoes. | 12 months
Reduction in 1st IMA from baseline to LOV | 6 months, 12 months
Number and type of Adverse Events | 6 months, 12 months
  Adverse events will be evaluated for their severity and frequency
Complications at surgery | 3 months
  Number and type of complications at surgery will be evaluated

OTHER OUTCOMES:
1st intermetatarsal forces at time of implantation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Elkahn Eliev, MD, Principal Investigator — MMC orthopedic department physician
Locations (1):
- MMC, Kfar Saba, Israel